CLINICAL TRIAL: NCT00581711
Title: Improving Otitis Media Care With EHR-based Clinical Decision Support and Feedback
Brief Title: Improving Otitis Media Care With Clinical Decision Support
Acronym: OMHIT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007-10-5555; 1R18HS017042-01 (AHRQ)
Record Dates: First submitted 2007-12-19; First posted 2007-12-28 (Estimated); Last update posted 2012-06-18 (Estimated); Status verified 2012-06

CONDITIONS: Otitis Media
Keywords: Electronic Health Record; Clinical Decision Support; Otitis Media
MeSH Terms: conditions — Otitis Media

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control (No Intervention): Usual Care
- HIT Intervention without feedback (Experimental): 3-Part Intervention: Training, Otitis Media Episode Grouper, Clinical Decision Support
  Interventions: Other: 3-Part Intervention
- HIT Intervention with feedback (Experimental): 4-Part Intervention: Training, Episode Grouper, Clinical Decision Support, and Physician Feedback.
  Interventions: Other: 4-Part Intervention
- Feedback only (Experimental): 1 part intervention: Physician Feedback
  Interventions: Other: 1-part intervention

INTERVENTIONS:
Other: 3-Part Intervention — A combination of training, an otitis media episode grouper, and clinical decision support.
  Arms: HIT Intervention without feedback
Other: 4-Part Intervention — A combination of clinician training, an otitis media episode grouper, clinical decision support, and feedback.
  Arms: HIT Intervention with feedback
Other: 1-part intervention — Provision of feedback on otitis media quality indicators
  Arms: Feedback only

SUMMARY:
This protocol will prospectively develop a new electronic health record (EHR)-based health information technology (IT) intervention that a) summarizes Otitis Media (OM) care into clinically meaningful episodes-of-care, b) provides clinical decision support based upon evidence-based guidelines to primary care and ENT physicians working within an integrated physician network that uses a common EHR, and c) tests the additive effects on quality and resource utilization of providing feedback to physicians.

DETAILED DESCRIPTION:
Context The high prevalence of Otitis Media (OM) and its enormous cost make it a prime target for cost-effective and evidence-based strategies for disease management.

Objectives

This protocol will prospectively develop a new electronic health record (EHR)-based health information technology (IT) intervention that a) summarizes OM care into clinically meaningful episodes-of-care, b) provides clinical decision support based upon evidence-based guidelines to primary care and ENT physicians working within an integrated physician network that uses a common EHR, and c) tests the additive effects on quality and resource utilization of providing feedback to physicians. The specific aims are:

Aim 1: To develop and pilot test the OM health IT intervention; Aim 2: To examine the overall effect of the health IT intervention and the independent contribution of physician feedback on quality of OM care (primary outcomes); Aim 3: To assess the effects of the intervention on the secondary outcomes of health care resource utilization and clinician adoption of the health IT.

Study Design/Settings/Participants A cluster randomized trial and multi-level statistical modeling will be used to estimate health IT intervention effects on study outcomes. The proposed project will be conducted in the Children's Hospital of Philadelphia's (CHOP) health care system. The heath IT intervention will be tested in the Pediatric Research Consortium (PeRC), which includes 28 primary care practices in the CHOP network, both urban and suburban, and the CHOP ENT clinical sites. Randomization and implementation of the intervention will occur at the practice level. Study outcomes of quality of care and resource utilization will be reported at the levels of the practice, individual practitioner, and episode-of-care (patient-level).

Study Measures Our main study measures include the quality of otitis media care provided during episodes of OM.

Our secondary outcomes include measurement of clinician adoption of the health IT intervention and resource use.

ELIGIBILITY:
Inclusion Criteria:

* All CHOP primary care pediatric and ENT practice sites are eligible for inclusion in this study. We expect 35,000 patients to receive care for otitis media by CHOP clinicians at these sites during the study period however, they are not the subjects of this research.

Exclusion Criteria:

* There are no exclusion criteria. All CHOP primary care pediatric and ENT sites are eligible for participation. Data for all clinicians providing OM care and data on all OM encounters will be included in our data set.

Ages: 2 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 55779 (Actual)
Dates: Start 2007-12; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Quality of otitis media care. | 18 Months

SECONDARY OUTCOMES:
Clinician adoption of intervention and Resource Utilization | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Christopher B Forrest, MD, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Forrest CB, Fiks AG, Bailey LC, Localio R, Grundmeier RW, Richards T, Karavite DJ, Elden L, Alessandrini EA. Improving adherence to otitis media guidelines with clinical decision support and physician feedback. Pediatrics. 2013 Apr;131(4):e1071-81. doi: 10.1542/peds.2012-1988. Epub 2013 Mar 11. PMID 23478860